CLINICAL TRIAL: NCT00929578
Title: Ascending-Dose, Double-Blind, Placebo-Controlled, Study of Intralesional Fluphenazine Hydrochloride for Psoriasis
Brief Title: Fluphenazine Hydrochloride for Psoriasis
Acronym: FP-CL2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: Immune Control (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FP-CL2
Record Dates: First submitted 2009-06-25; First posted 2009-06-29 (Estimated); Results first posted 2016-08-02 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Psoriasis
Keywords: Psoriasis; T-lymphocytes; Fluphenazine
MeSH Terms: conditions — Psoriasis | interventions — Fluphenazine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): The sterile placebo: Bacteriostatic Sodium Chloride for Injection.
  Interventions: Drug: Placebo
- Fluphenazine (Active Comparator): This will be an ascending dose study with the first cohort of 5 subjects dosed at 100 µg/mL, followed by cohorts at 500 and 2500 µg/mL. Dosing will be on Days 0, 7 and 14 and will consist of 5, or 10, 100 µL injections into the psoriatic lesion. The number of injections will depend on the lesion size. As this is a vehicle controlled study, subjects will receive intralesional injections of both drug and placebo, each into a separate target plaque, in a randomized fashion.
  Interventions: Drug: Fluphenazine

INTERVENTIONS:
Drug: Fluphenazine — Intralesional injection of Fluphenazine
  Other Names: FP-CL2
  Arms: Fluphenazine
Drug: Placebo — Intralesional injection of placebo
  Other Names: Bacteriostatic Sodium Chloride
  Arms: Placebo

SUMMARY:
The objective of this study is to assess the safety and biologic activity of intralesional injection of fluphenazine in adult subjects with psoriasis.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, bilateral, ascending dose study.

In vitro, fluphenazine has been shown to suppress growth of proliferating T-lymphocytes. Fluphenazine would be expected to also suppress growth of proliferating T-lymphocytes in psoriatic plaques.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 to 65 years of age with psoriasis, in general good health as determined by the Principal Investigator based upon the results of medical history, laboratory profile, and physical examination
* Must have symmetric target lesions 2-4 cm in diameter on each side of the body (e.g., thighs) with baseline Target Lesion Score (TLS) of 6 or higher (scale of 0-12) for each target
* Women are eligible to participate in the study if they meet one of the following criteria:

  * Women who are postmenopausal (for at least one year), sterile, or hysterectomized
  * Women of childbearing potential must undergo monthly pregnancy testing during the study and agree to use two of the following methods of contraception throughout the study and for 60 days after the last dose of study drug:

    * Oral contraceptives
    * Transdermal contraceptives
    * Injectable or implantable methods
    * Intrauterine devices
    * Barrier methods (diaphragm with spermicide, condom with spermicide)

(Abstinence and Tubal Ligation are also considered a form of Birth control.)

Exclusion Criteria:

* Patient is not asymptomatic and has major ailments on screening exam.
* Infliximab (Remicade®) or alefacept (Amevive®) within the past 6 months (24 weeks)
* Etanercept (Enbrel®), efalizumab (Raptiva™), adalimumab (Humira®) or other tumor necrosis factor (TNF)-alpha inhibitor within the past 3 months (12 weeks)
* Other systemic psoriasis therapies (e.g., methotrexate, cyclosporine, acitretin) or oral psoralen with ultraviolet A (PUVA) within the past 4 weeks
* ultraviolet B (UVB) or topical therapy (other than over-the-counter (OTC) moisturizers and shampoos) within the past 2 weeks (including topical corticosteroids, vitamin A and D analogues) with the exception of betamethasone valerate lotion (0.01%) for treatment of scalp lesions, and triamcinolone cream (0.1%) for lesions at least 3 inches away from the target lesions
* Receipt of an investigation agent within the past 4 weeks
* Systemic corticosteroid therapy
* Inability to understand consent or comply with protocol (patients will be asked if they understand or have any questions)
* Pregnancy, lactation, or unwillingness to use adequate birth control during the study
* Impaired hepatic function
* Known HIV/AIDS, hepatitis B/C
* Blood dyscrasia
* Epilepsy
* Tardive dyskinesia
* Excessive alcohol consumption (drinking more than two drinks per day on average for men or more than one drink per day on average for women)
* Use of phenothiazine antipsychotics or anticholinergics
* Current use of selective serotonin reuptake inhibitor (SSRI), tricyclic, or norepinephrine reuptake inhibitor antidepressants or use within 6 weeks of beginning the study
* Concurrent use of anti-seizure drugs, with the exception of gabapentin for treatment of neuropathy
* Known allergy to fluphenazine or other phenothiazines, sesame oil or sesame seeds
* Known allergy to parabens, para-aminobenzoate (PABA) or benzyl alcohol
* Clinically significant and uncontrolled cardiovascular disease
* corrected QT interval (QTc) > 450 msec, or evidence of a clinically significant dysrhythmia on ECG
* Operator of heavy machinery
* Pheochromocytoma
* Clinically significant mitral valve disease
* History of breast cancer
* History of seizure disorder
* Occupational exposure to organophosphate insecticides
* Parkinson's disease and other related movement disorders
* Screening Lab abnormalities including:

  * Serum Asparate transaminase (AST) or Alanine transaminase (ALT) > 2.5 upper limits of normal
  * Creatinine ≥ 1.6 mg/dL
  * Bilirubin ≥ 1.5 mg/dL
  * White blood cell (WBC) count < 3 x 10^9 /L
  * Platelets < 100 x 10^9/L
  * Hemoglobin < 10 g/dL in females or < 12g/dL in males
  * Glucose ≥ 200 mg/dL
  * Fasting blood sugar ≥ 126 mg/dL
* Concurrent use of drugs listed in Appendix E of protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-11; Primary Completion 2010-11 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alice B. Gottlieb, M.D., PhD., Principal Investigator — Tufts Medical Center, Department of Dermatology
Locations (2):
- United States (2):
  - Tufts Medical Center, Department of Dermatology, Boston, Massachusetts
  - Robert Wood Johnson Medical School, Psoriasis Center of Excellence, New Brunswick, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gupta MA, Guptat AK. The use of antidepressant drugs in dermatology. J Eur Acad Dermatol Venereol. 2001 Nov;15(6):512-8. doi: 10.1046/j.1468-3083.2001.00278.x. PMID 11843209

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from a dermatology clinic of a tertiary care medical center. Recruitment dates from Oct 2008 to Sep 2010.
Groups:
- All Study Participants: The sterile placebo: Bacteriostatic Sodium Chloride for Injection. Same subject will also receive dose in other arm of fluphenazine. This will be an ascending dose study with the first cohort of 5 subjects dosed at 100 µg/mL, followed by cohorts at 500 and 2500 µg/mL. Dosing will be on Days 0, 7 and 14 and will consist of 5, or 10, 100 µL injections into the psoriatic lesion. The number of injections will depend on the lesion size. As this is a vehicle controlled study, subjects will receive intralesional injections of both drug and placebo, each into a separate target plaque, in a randomized fashion.
Period: Overall Study
Arm/Group | All Study Participants
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants - Fluphenazine: This will be an ascending dose study with the first cohort of 5 subjects dosed at 100 µg/mL, followed by cohorts at 500 and 2500 µg/mL. Dosing will be on Days 0, 7 and 14 and will consist of 5, or 10, 100 µL injections into the psoriatic lesion. The number of injections will depend on the lesion size. As this is a vehicle controlled study, subjects will receive intralesional injections of both drug and placebo, each into a separate target plaque, in a randomized fashion.
Arm/Group | All Study Participants - Fluphenazine
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Target Lesion Scoring Evaluated at Baseline and 4 Weeks
Description: Actual change in target lesion score comparing 4 week score with baseline score. Improvement is positive, worsening is negative. Target lesions scores range from 0 (no disease) to 12 (severe disease), and are scored based on the sum of erythema (0-4), induration (0-4) and scale (0-4) scores.
Time Frame: 4 weeks
Population: All participants who successfully were enrolled.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Fluphenazine
Number analyzed (Participants) | 15 | 15
units on a scale | -1.4 (1.5) | -1.4 (1.8)

2. Secondary Outcome: Change in the Target Lesion Visual Analog Scale (VAS) Score for Pruritus Evaluated at Baseline and 4 Weeks
Description: Visual Analog Scale (VAS) score for pruritus. Subjective measurement of pruritus on an analog scale with a single mark denoting self-perceived pruritus: Minimum 0mm for no itch, Maximum 100mm for worst itch imaginable. Scores are measured in millimeters. This secondary outcome is a percentage improvement from baseline score for pruritus. Improvement is negative, worsening is positive.
Time Frame: 4 weeks
Population: Participants who completed entire trial.
Measure: Mean (Standard Deviation); unit: percentage of baseline pruritus
Arm/Group | Placebo | Fluphenazine
Number analyzed (Participants) | 15 | 15
percentage of baseline pruritus | 0.86 (15.0) | -2.16 (22.9)

3. Secondary Outcome: Safety Outcome Measures
Description: adverse events will be recorded and monitored. Adverse events will be noted in a separate chart.
Time Frame: 8 weeks
Population: All participants who completed enrollment.
Measure: Number; unit: All Study Participant
Groups:
- All Study Participants: Participants who experienced at least one adverse event.
Arm/Group | All Study Participants
Number analyzed (Participants) | 15
All Study Participant | 12

4. Secondary Outcome: Fluphenazine Serum Levels Measured at Baseline, 2 Hours Post Dose and 1 Week Post Dose.
Description: Number of participants with fluphenazine serum levels > 0.200ng/ml, at baseline, 2 hours post dose and 1 week post dose.
Time Frame: 1 week
Population: All participants who were enrolled and completed baseline and week 1 were included.
Measure: Number; unit: participants
Groups:
- Baseline: Number of participants with fluphenazine serum levels > 0.200ng/ml at baseline
- 2 Hours Post Dose: Number of participants with fluphenazine serum levels > 0.200ng/ml, 2 hours after administration
- 1 Week Post Dose: Participants with fluphenazine serum levels > 0.200ng/ml
Arm/Group | Baseline | 2 Hours Post Dose | 1 Week Post Dose
Number analyzed (Participants) | 15 | 15 | 15
participants | 0 | 2 | 2

ADVERSE EVENTS:
Time Frame: 1 year, 10 months
Groups:
- All Study Participants: This will be an ascending dose study with the first cohort of 5 subjects dosed at 100 µg/mL, followed by cohorts at 500 and 2500 µg/mL. Dosing will be on Days 0, 7 and 14 and will consist of 5, or 10, 100 µL injections into the psoriatic lesion. The number of injections will depend on the lesion size. As this is a vehicle controlled study, subjects will receive intralesional injections of both drug and placebo, each into a separate target plaque, in a randomized fashion. All participants received medication, as the study was a split study, and subjects received placebo on one side and injection of fluphenazine on other side
Arm/Group | All Study Participants
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 12/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Participants (N=15)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Self limited Upper Respiratory Infection
Difficulty Sleeping (General disorders) | 2 (2)
Fatigue (General disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Xerosis (Skin and subcutaneous tissue disorders) | 1 (1)
Dry Eyes (Eye disorders) | 1 (1)
Injection Site Pain (Skin and subcutaneous tissue disorders) | 2 (2)
Sprained Medial Collateral Ligament (Musculoskeletal and connective tissue disorders) | 1 (1)
Nighttime Sweats (Skin and subcutaneous tissue disorders) | 1 (1)
Bruise, Upper left arm (Skin and subcutaneous tissue disorders) | 1 (1)
Nightmares (Psychiatric disorders) | 1 (1)
Dry mouth (General disorders) | 1 (1)
Gout (Musculoskeletal and connective tissue disorders) | 1 (1)
Blisters (Skin and subcutaneous tissue disorders) | 1 (1)
Ankle Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Unusual dreams (General disorders) | 2 (2)
Abrasion (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No